CLINICAL TRIAL: NCT00255190
Title: A Phase 3, Open-Label Study to Assess the Long-Term Safety of Dexlansoprazole MR (60 mg QD and 90 mg QD)
Brief Title: Safety and Quality of Life Study of Dexlansoprazole Modified Release Formulation to Treat Heartburn
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T-GI04-088; U1111-1114-0151 (Registry Identifier: WHO)
Record Dates: First submitted 2005-11-15; First posted 2005-11-17 (Estimated); Results first posted 2009-08-12 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2011-04

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: Gastroesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Dexlansoprazole; Lansoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexlansoprazole MR 60 mg QD (Experimental)
  Interventions: Drug: Dexlansoprazole MR
- Dexlansoprazole MR 90 mg QD (Experimental)
  Interventions: Drug: Dexlansoprazole MR

INTERVENTIONS:
Drug: Dexlansoprazole MR — Dexlansoprazole MR 60 mg, capsules, orally, once daily for up to 12 months.
  Other Names: TAK-390MR; Kapidex; Dexilant
  Arms: Dexlansoprazole MR 60 mg QD
Drug: Dexlansoprazole MR — Dexlansoprazole MR 90 mg, capsules, orally, once daily for up to 12 months.
  Other Names: TAK-390MR; Kapidex; Dexilant
  Arms: Dexlansoprazole MR 90 mg QD

SUMMARY:
The purpose of this study is to determine the long-term safety profile of daily treatment with dexlansoprazole MR in subjects with gastroesophageal reflux disease.

DETAILED DESCRIPTION:
This open-label study is intended to determine the long-term safety profile of dexlansoprazole MR over 12 months of dosing with 60 mg once-daily (QD) or 90 mg QD in subjects with gastroesophageal reflux disease (GERD), including those with esophageal erosions.

Prior to a protocol amendment, 300 subjects successfully completed one of the symptomatic nonerosive gastroesophageal reflux studies T-GD04-082 (NCT00251745) or T-GD04-083 (NCT00251758) in which they were randomly assigned to receive placebo or dexlansoprazole MR 60 or 90 mg QD. Subjects who were enrolled from one of these symptomatic GERD studies were randomly assigned in a 1:1 ratio to receive either dexlansoprazole MR 60 or 90 mg QD in this long-term study.

After implementation of protocol amendment #4, an additional 300 subjects with gastroesophageal reflux disease including those with erosive esophagitis will be enrolled and treated with dexlansoprazole MR 90 mg QD for 12 months.

Approximately 200 study sites in the U.S. will participate.

For all analyses involving visits during treatment from subjects enrolled prior to protocol amendment #4, baseline refers to pretreatment to Study T-GD04-082 (NCT00251745) or T-GD04-083 (NCT00251758). For subjects enrolled under protocol amendment #4, baseline is based on screening or predosing measurement.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have successfully completed either T-GD04-082 (NCT00251745) or T-GD04-083 (NCT00251758) or have a diagnosis of gastroesophageal reflux disease with or without erosive esophagitis.

Exclusion Criteria:

* Any condition that may require inpatient surgery during the course of the study.
* Use of prescription or non-prescription proton pump inhibitors, histamine (H2) receptor antagonists, sucralfate, misoprostol or prokinetics throughout the study.
* Use of antacids [except for study supplied Gelusil®].
* Subjects using drugs with significant anticholinergic effects such as tricyclics who cannot stay on a stable dose for 4 weeks prior to dosing and throughout the study.
* Evidence of uncontrolled systemic disease.
* Allergy to any proton pump inhibitor including Prilosec, Nexium, Prevacid, or others, any component of dexlansoprazole MR, or Gelusil/antacid.
* Need to take blood thinners.
* Need to take more than 12 doses of non-steroidal anti-inflammatory drugs per month.
* Had cancer (except basal cell cancer of the skin) within 3 years prior to screening.
* Has other esophageal disease including Barrett's esophagus or strictures requiring dilation.
* Has had radiation or cryotherapy to the esophagus.
* Has active gastric or duodenal ulcers within 4 weeks of starting study drug.
* Has a history of hypersecretory conditions such as Zollinger Ellison Syndrome.
* History of alcohol abuse.
* Has acquired immunodeficiency syndrome.
* Has had acute upper gastrointestinal bleeding within 4 weeks of endoscopy.
* Received a blood product transfusion within 3 months of taking the first dose of study drug.
* Has previously participated in another dexlansoprazole MR long-term treatment clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 591 (Actual)
Dates: Start 2006-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (181):
- United States (181):
  - Alabaster, Alabama
  - Anniston, Alabama
  - Birmingham, Alabama
  - Hueytown, Alabama
  - Huntsville, Alabama
  - Mobile, Alabama
  - Tallassee, Alabama
  - Tuscaloosa, Alabama
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - North Little Rock, Arkansas
  - Anaheim, California
  - Azusa, California
  - Carmichael, California
  - Chula Vista, California
  - Cypress, California
  - Fresno, California
  - Fullerton, California
  - Garden Grove, California
  - Irvine, California
  - Lancaster, California
  - Long Beach, California
  - Los Angeles, California
  - Mission Hills, California
  - Modesto, California
  - Newport Beach, California
  - Oakland, California
  - Orange, California
  - Palm Springs, California
  - Pasadena, California
  - Redwood City, California
  - San Diego, California
  - San Luis Obispo, California
  - Santa Maria, California
  - Boulder, Colorado
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Littleton, Colorado
  - Lone Tree, Colorado
  - Longmont, Colorado
  - Wheat Ridge, Colorado
  - Bristol, Connecticut
  - Waterbury, Connecticut
  - Newark, Delaware
  - Boynton Beach, Florida
  - Fort Myers, Florida
  - Jacksonville, Florida
  - Jupiter, Florida
  - Kissimmee, Florida
  - Lakeland, Florida
  - Miami, Florida
  - Naples, Florida
  - New Port Richey, Florida
  - New Smyrna Beach, Florida
  - Ocala, Florida
  - Pembroke Pines, Florida
  - Port Orange, Florida
  - Sarasota, Florida
  - St. Petersburg, Florida
  - Zephyrhills, Florida
  - Atlanta, Georgia
  - Honolulu, Hawaii
  - Arlington Heights, Illinois
  - Champaign, Illinois
  - Chicago, Illinois
  - Hines, Illinois
  - Moline, Illinois
  - North Chicago, Illinois
  - Oak Forest, Illinois
  - Oak Park, Illinois
  - Rockford, Illinois
  - Springfield, Illinois
  - Evansville, Indiana
  - Indianapolis, Indiana
  - Newburgh, Indiana
  - Clive, Iowa
  - Davenport, Iowa
  - Dubuque, Iowa
  - Kansas City, Kansas
  - Newton, Kansas
  - Shawnee Mission, Kansas
  - Topeka, Kansas
  - Wichita, Kansas
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Baton Rouge, Louisiana
  - Metairie, Louisiana
  - Shreveport, Louisiana
  - Chevy Chase, Maryland
  - Hollywood, Maryland
  - Lutherville, Maryland
  - Prince Frederick, Maryland
  - Troy, Michigan
  - Chaska, Minnesota
  - Jackson, Mississippi
  - Jefferson City, Missouri
  - Kansas City, Missouri
  - Mexico, Missouri
  - St Louis, Missouri
  - Washington, Missouri
  - Missoula, Montana
  - Omaha, Nebraska
  - Pahrump, Nevada
  - Egg Harbor, New Jersey
  - New Brunswick, New Jersey
  - Albuquerque, New Mexico
  - Binghamton, New York
  - Brooklyn, New York
  - Great Neck, New York
  - Rochester, New York
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Elkin, North Carolina
  - Greensboro, North Carolina
  - Harrisburg, North Carolina
  - Hickory, North Carolina
  - High Point, North Carolina
  - Raleigh, North Carolina
  - Salisbury, North Carolina
  - Statesville, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Bismarck, North Dakota
  - Akron, Ohio
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Dayton, Ohio
  - Mayfield Heights, Ohio
  - Mogadore, Ohio
  - Warren, Ohio
  - Oklahoma City, Oklahoma
  - Medford, Oregon
  - Portland, Oregon
  - Beaver Falls, Pennsylvania
  - Duncansville, Pennsylvania
  - Lansdale, Pennsylvania
  - Philadelphia, Pennsylvania
  - Warwick, Rhode Island
  - Anderson, South Carolina
  - Mt. Pleasant, South Carolina
  - Sioux Falls, South Dakota
  - Bristol, Tennessee
  - Chattanooga, Tennessee
  - Germantown, Tennessee
  - Hermitage, Tennessee
  - Jackson, Tennessee
  - Johnson City, Tennessee
  - Kingsport, Tennessee
  - Nashville, Tennessee
  - Amarillo, Texas
  - Austin, Texas
  - Beaumont, Texas
  - Bryan, Texas
  - Conroe, Texas
  - Corsicana, Texas
  - Dallas, Texas
  - El Paso, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Odessa, Texas
  - Pharr, Texas
  - San Antonio, Texas
  - Seguin, Texas
  - Tyler, Texas
  - Bountiful, Utah
  - Ogden, Utah
  - Salt Lake City, Utah
  - West Jordan, Utah
  - Charlottesville, Virginia
  - Chesapeake, Virginia
  - Danville, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
  - Bellevue, Washington
  - Lakewood, Washington
  - Spokane, Washington
  - Tacoma, Washington
  - Milwaukee, Wisconsin
  - Monroe, Wisconsin

REFERENCES:
- [Result] Friedlander EA, Pallentino J, Miller SK, VanBeuge SS. The evolution of proton pump inhibitors for the treatment of gastroesophageal reflux disease. J Am Acad Nurse Pract. 2010 Dec;22(12):674-83. doi: 10.1111/j.1745-7599.2010.00578.x. Epub 2010 Nov 24. PMID 21129076
- [Result] Dabholkar AH, Han C, Paris MM, Perez MC, Atkinson SN, Peura DA. The 12-month safety profile of dexlansoprazole, a proton pump inhibitor with a dual delayed release formulation, in patients with gastro-oesophageal reflux disease. Aliment Pharmacol Ther. 2011 Feb;33(3):366-77. doi: 10.1111/j.1365-2036.2010.04519.x. Epub 2010 Nov 30. PMID 21118280
- [Result] Peura DA, Metz DC, Dabholkar AH, Paris MM, Yu P, Atkinson SN. Safety profile of dexlansoprazole MR, a proton pump inhibitor with a novel dual delayed release formulation: global clinical trial experience. Aliment Pharmacol Ther. 2009 Nov 15;30(10):1010-21. doi: 10.1111/j.1365-2036.2009.04137.x. Epub 2009 Sep 4. PMID 19735233
- See also: Dexilant Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=9efb34b3-fb69-4190-a2be-a90b8cb94e25&filetypecode=DEXILANTPI

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 104 sites in the United States from 07 January 2006 to 25 June 2008.
Pre-assignment Details: At screening, subjects completed a Patient Assessment of Upper Gastrointestinal Disorders Quality-of-Life Index (PAGI-QOL) and Patient Assessment of Upper Gastrointestinal Disorders-Symptom Severity Index (PAGI-SYM) questionnaires before enrollment in Dexlansoprazole Modified Release (MR) 60 mg or 90 mg once daily (QD) treatment groups.
Groups:
- Dexlansoprazole MR 60 mg QD: Dexlansoprazole MR 60 mg, orally, once daily for up to 12 months
- Dexlansoprazole MR 90 mg QD: Dexlansoprazole MR 90 mg, orally, once daily for up to 12 months
Period: Overall Study
Arm/Group | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Started | 153 | 438
Completed | 103 | 281
Not Completed | 50 | 157
Not completed — Adverse Event | 17 | 36
Not completed — Protocol Violation | 2 | 2
Not completed — Lost to Follow-up | 10 | 27
Not completed — Withdrew Consent | 17 | 48
Not completed — Inclusion/Exclusion criteria not met | 0 | 1
Not completed — Erosive esophagitis not healed | 0 | 20
Not completed — Various | 4 | 23

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD | Total
Number analyzed (Participants) | 153 | 438 | 591
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (13.78) | 49.0 (13.50) | 48.7 (13.57)
Age, Customized [Number; unit: subjects]
  <45 years | 65 | 158 | 223
  45 to <65 years | 71 | 237 | 308
  ≥65 years | 17 | 43 | 60
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 283 | 388
  Male | 48 | 155 | 203
Race/Ethnicity, Customized [Number; unit: subjects]
  American Indian or Alaska Native | 3 | 8 | 11
  Asian | 6 | 14 | 20
  Black of African Heritage | 18 | 44 | 62
  White | 126 | 366 | 492
  Multiracial | 0 | 6 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 64 | 88
  Not Hispanic or Latino | 129 | 374 | 503
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: subjects]
  United States | 153 | 438 | 591

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to Month 12 for Hemoglobin Values
Time Frame: Baseline and Month 12
Population: All subjects who received at least 1 dose of study drug are included in safety analyses. For changes from baseline, a subject had to have a baseline value and a Month 12 value to be included in the summary of a specific parameter.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Number analyzed (Participants) | 88 | 228
g/dL | -0.29 (0.873) | -0.05 (0.959)
Statistical Analysis 1: Comparison: Dexlansoprazole MR 60 mg QD vs Dexlansoprazole MR 90 mg QD; Test type: Superiority or Other; p = 0.042, ANOVA — Statistical significance was determined at 0.05 level. All statistical tests were two-sided and the p-values were rounded to 3 decimal places prior to determining statistical significance

2. Primary Outcome: Mean Change From Baseline to Month 12 for Hematocrit Values
Description: Hematocrit measurement percent is the absolute difference in Hematocrit values, and not percentage difference.
Time Frame: Baseline and Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Number analyzed (Participants) | 88 | 228
percentage | -1.98 (2.573) | -0.93 (3.156)
Statistical Analysis 1: Comparison: Dexlansoprazole MR 60 mg QD vs Dexlansoprazole MR 90 mg QD; Test type: Superiority or Other; p = 0.006, ANOVA — [p-value comment as in outcome 1, analysis 1]

3. Secondary Outcome: Mean Change From Baseline to Month 1 for PAGI-QOL Total Score
Description: Mean overall composite Quality of Life (QOL) score changes were computed in response to 30 questions, each scored 0 (lowest QOL) to 5 (highest QOL). Positive changes from baseline indicate improved QOL.
Time Frame: Baseline and Month 1
Population: All subjects who received at least 1 dose of study drug and had a value for ≥1 subscale at both baseline and after Day 1 were included in the Patient Assessment of Upper Gastrointestinal Disorders (PAGI) analyses.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Number analyzed (Participants) | 143 | 406
score on a scale | 0.54 (0.718) | 0.54 (0.735)
Statistical Analysis 1: Comparison: Dexlansoprazole MR 60 mg QD vs Dexlansoprazole MR 90 mg QD; Test type: Superiority or Other; p = 0.204, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Comparisons were made using a one-way analysis of covariance (ANCOVA) model with treatment as the factor and baseline score as the covariate

4. Secondary Outcome: Mean Change From Baseline to Month 3 for PAGI-QOL Total Score
Description: Mean overall composite QOL score changes were computed in response to 30 questions, each scored 0 (lowest QOL) to 5 (highest QOL). Positive changes from baseline indicate improved QOL.
Time Frame: Baseline and Month 3
Population: All subjects who received at least 1 dose of study drug and had a value for ≥1 subscale at both baseline and after Day 1 were included in the PAGI analyses.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Number analyzed (Participants) | 130 | 377
score on a scale | 0.61 (0.827) | 0.56 (0.754)
Statistical Analysis 1: Comparison: Dexlansoprazole MR 60 mg QD vs Dexlansoprazole MR 90 mg QD; Test type: Superiority or Other; p = 0.109, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Comparisons were made using an ANCOVA model with treatment as the factor and baseline score as the covariate

5. Primary Outcome: Mean Change From Baseline to Month 12 for Red Blood Cell Count Values
Time Frame: Baseline and Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Red Blood Cell count x10 to the 6/μL
Arm/Group | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Number analyzed (Participants) | 88 | 228
Red Blood Cell count x10 to the 6/μL | -0.31 (0.271) | -0.11 (0.349)
Statistical Analysis 1: Comparison: Dexlansoprazole MR 60 mg QD vs Dexlansoprazole MR 90 mg QD; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 1, analysis 1]

6. Primary Outcome: Mean Change From Baseline to Month 12 for Mean Corpuscular Hemoglobin Concentration Values
Time Frame: Baseline and Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Number analyzed (Participants) | 88 | 228
g/dL | 0.67 (1.428) | 0.56 (1.277)
Statistical Analysis 1: Comparison: Dexlansoprazole MR 60 mg QD vs Dexlansoprazole MR 90 mg QD; Test type: Superiority or Other; p = 0.494, ANOVA — [p-value comment as in outcome 1, analysis 1]

7. Primary Outcome: Mean Change From Baseline to Month 12 for Platelet Count Values
Time Frame: Baseline and Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Platelet Count x10 to the 3/mcL
Arm/Group | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Number analyzed (Participants) | 88 | 224
Platelet Count x10 to the 3/mcL | -12.7 (36.24) | -1.9 (39.31)
Statistical Analysis 1: Comparison: Dexlansoprazole MR 60 mg QD vs Dexlansoprazole MR 90 mg QD; Test type: Superiority or Other; p = 0.026, ANOVA — [p-value comment as in outcome 1, analysis 1]

8. Primary Outcome: Mean Change From Baseline to Month 12 for White Blood Cell Count Values
Time Frame: Baseline and Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: White Blood Cell count x10 to the 3/mcL
Arm/Group | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Number analyzed (Participants) | 88 | 228
White Blood Cell count x10 to the 3/mcL | -0.20 (1.610) | 0.04 (1.624)
Statistical Analysis 1: Comparison: Dexlansoprazole MR 60 mg QD vs Dexlansoprazole MR 90 mg QD; Test type: Superiority or Other; p = 0.220, ANOVA — [p-value comment as in outcome 1, analysis 1]

9. Primary Outcome: Mean Change From Baseline to Month 12 for Blood Urea Nitrogen Values
Time Frame: Baseline and Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Number analyzed (Participants) | 89 | 232
mg/dL | 0.1 (4.58) | 0.0 (4.03)
Statistical Analysis 1: Comparison: Dexlansoprazole MR 60 mg QD vs Dexlansoprazole MR 90 mg QD; Test type: Superiority or Other; p = 0.843, ANOVA — [p-value comment as in outcome 1, analysis 1]

10. Primary Outcome: Mean Change From Baseline to Month 12 for Creatinine Values
Time Frame: Baseline and Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Number analyzed (Participants) | 89 | 232
mg/dL | -0.04 (0.323) | -0.04 (0.111)
Statistical Analysis 1: Comparison: Dexlansoprazole MR 60 mg QD vs Dexlansoprazole MR 90 mg QD; Test type: Superiority or Other; p = 0.923, ANOVA — [p-value comment as in outcome 1, analysis 1]

11. Primary Outcome: Mean Change From Baseline to Month 12 for Calcium Values
Time Frame: Baseline and Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Number analyzed (Participants) | 89 | 232
mg/dL | -0.25 (0.421) | -0.04 (0.443)
Statistical Analysis 1: Comparison: Dexlansoprazole MR 60 mg QD vs Dexlansoprazole MR 90 mg QD; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 1, analysis 1]

12. Primary Outcome: Mean Change From Baseline to Month 12 for Inorganic Phosphorus Values
Time Frame: Baseline and Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Number analyzed (Participants) | 89 | 231
mg/dL | 0.09 (0.613) | 0.06 (0.730)
Statistical Analysis 1: Comparison: Dexlansoprazole MR 60 mg QD vs Dexlansoprazole MR 90 mg QD; Test type: Superiority or Other; p = 0.758, ANOVA — [p-value comment as in outcome 1, analysis 1]

13. Primary Outcome: Mean Change From Baseline to Month 12 for Total Bilirubin Values
Time Frame: Baseline and Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Number analyzed (Participants) | 89 | 231
mg/dL | -0.02 (0.166) | -0.01 (0.170)
Statistical Analysis 1: Comparison: Dexlansoprazole MR 60 mg QD vs Dexlansoprazole MR 90 mg QD; Test type: Superiority or Other; p = 0.737, ANOVA — [p-value comment as in outcome 1, analysis 1]

14. Primary Outcome: Mean Change From Baseline to Month 12 for Alkaline Phosphatase Values
Time Frame: Baseline and Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Number analyzed (Participants) | 89 | 231
U/L | 0.4 (11.59) | -0.4 (14.69)
Statistical Analysis 1: Comparison: Dexlansoprazole MR 60 mg QD vs Dexlansoprazole MR 90 mg QD; Test type: Superiority or Other; p = 0.673, ANOVA — [p-value comment as in outcome 1, analysis 1]

15. Primary Outcome: Mean Change From Baseline to Month 12 for Aspartate Aminotransferase Values
Time Frame: Baseline and Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Number analyzed (Participants) | 88 | 221
U/L | 0.9 (7.81) | 0.6 (10.14)
Statistical Analysis 1: Comparison: Dexlansoprazole MR 60 mg QD vs Dexlansoprazole MR 90 mg QD; Test type: Superiority or Other; p = 0.817, ANOVA — [p-value comment as in outcome 1, analysis 1]

16. Primary Outcome: Mean Change From Baseline to Month 12 for Alanine Aminotransferase Values
Time Frame: Baseline and Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Number analyzed (Participants) | 89 | 226
U/L | 1.6 (10.43) | 0.5 (17.43)
Statistical Analysis 1: Comparison: Dexlansoprazole MR 60 mg QD vs Dexlansoprazole MR 90 mg QD; Test type: Superiority or Other; p = 0.601, ANOVA — [p-value comment as in outcome 1, analysis 1]

17. Primary Outcome: Mean Change From Baseline to Month 12 for Serum Gastrin Levels
Time Frame: Baseline and Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Number analyzed (Participants) | 81 | 208
pg/mL | 155.8 (189.67) | 115.4 (156.32)
Statistical Analysis 1: Comparison: Dexlansoprazole MR 60 mg QD vs Dexlansoprazole MR 90 mg QD; Test type: Superiority or Other; p = 0.065, ANOVA — [p-value comment as in outcome 1, analysis 1]

18. Primary Outcome: Mean Change From Baseline to Month 12 for Systolic Blood Pressure
Time Frame: Baseline and Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Number analyzed (Participants) | 88 | 237
mm Hg | 3.8 (15.37) | 1.9 (14.91)
Statistical Analysis 1: Comparison: Dexlansoprazole MR 60 mg QD vs Dexlansoprazole MR 90 mg QD; Test type: Superiority or Other; p = 0.319, ANOVA — [p-value comment as in outcome 1, analysis 1]

19. Primary Outcome: Mean Change From Baseline to Month 12 for Diastolic Blood Pressure
Time Frame: Baseline and Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Number analyzed (Participants) | 88 | 237
mm Hg | 4.0 (9.53) | 0.6 (11.03)
Statistical Analysis 1: Comparison: Dexlansoprazole MR 60 mg QD vs Dexlansoprazole MR 90 mg QD; Test type: Superiority or Other; p = 0.011, ANOVA — [p-value comment as in outcome 1, analysis 1]

20. Primary Outcome: Mean Change From Baseline to Month 12 for Pulse Rate
Time Frame: Baseline and Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Number analyzed (Participants) | 88 | 237
beats per minute | 0.5 (10.11) | -1.3 (11.87)
Statistical Analysis 1: Comparison: Dexlansoprazole MR 60 mg QD vs Dexlansoprazole MR 90 mg QD; Test type: Superiority or Other; p = 0.207, ANOVA — [p-value comment as in outcome 1, analysis 1]

21. Secondary Outcome: Mean Change From Baseline to Month 6 for PAGI-QOL Total Score
Description: as for outcome 4
Time Frame: Baseline and Month 6
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Number analyzed (Participants) | 119 | 329
score on a scale | 0.58 (0.792) | 0.56 (0.758)
Statistical Analysis 1: Comparison: Dexlansoprazole MR 60 mg QD vs Dexlansoprazole MR 90 mg QD; Test type: Superiority or Other; p = 0.286, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Comparisons were made using an ANCOVA model with treatment as the factor and baseline score as the covariate

22. Secondary Outcome: Mean Change From Baseline to Month 9 for PAGI-QOL Total Score
Description: as for outcome 4
Time Frame: Baseline and Month 9
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Number analyzed (Participants) | 110 | 303
score on a scale | 0.64 (0.757) | 0.60 (0.811)
Statistical Analysis 1: Comparison: Dexlansoprazole MR 60 mg QD vs Dexlansoprazole MR 90 mg QD; Test type: Superiority or Other; p = 0.102, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Comparisons were made using an ANCOVA model with treatment as the factor and baseline score as the covariate

23. Secondary Outcome: Mean Change From Baseline to Month 12 for PAGI-QOL Total Score
Description: as for outcome 4
Time Frame: Baseline and Month 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Number analyzed (Participants) | 95 | 244
score on a scale | 0.56 (0.725) | 0.61 (0.809)
Statistical Analysis 1: Comparison: Dexlansoprazole MR 60 mg QD vs Dexlansoprazole MR 90 mg QD; Test type: Superiority or Other; p = 0.656, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Comparisons were made using an ANCOVA model with treatment as the factor and baseline score as the covariate

24. Secondary Outcome: Mean Change From Baseline to Month 1 for PAGI-SYM Total Score
Description: Mean overall composite symptom-severity score changes were computed in response to 20 questions, each scored 0 (no symptoms) to 5 (most severe symptoms). Negative changes from baseline indicate improvement in symptoms (decrease in severity).
Time Frame: Baseline and Month 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Number analyzed (Participants) | 143 | 394
score on a scale | -0.95 (0.876) | -0.85 (0.874)
Statistical Analysis 1: Comparison: Dexlansoprazole MR 60 mg QD vs Dexlansoprazole MR 90 mg QD; Test type: Superiority or Other; p = 0.176, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Comparisons were made using an ANCOVA model with treatment as the factor and baseline score as the covariate

25. Secondary Outcome: Mean Change From Baseline to Month 3 for PAGI-SYM Total Score
Description: as for outcome 24
Time Frame: Baseline and Month 3
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Number analyzed (Participants) | 130 | 364
score on a scale | -1.09 (0.913) | -0.91 (0.896)
Statistical Analysis 1: Comparison: Dexlansoprazole MR 60 mg QD vs Dexlansoprazole MR 90 mg QD; Test type: Superiority or Other; p = 0.030, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Comparisons were made using an ANCOVA model with treatment as the factor and baseline score as the covariate

26. Secondary Outcome: Mean Change From Baseline to Month 6 for PAGI-SYM Total Score
Description: as for outcome 24
Time Frame: Baseline and Month 6
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Number analyzed (Participants) | 119 | 318
score on a scale | -1.05 (0.885) | -0.93 (0.856)
Statistical Analysis 1: Comparison: Dexlansoprazole MR 60 mg QD vs Dexlansoprazole MR 90 mg QD; Test type: Superiority or Other; p = 0.243, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Comparisons were made using an ANCOVA model with treatment as the factor and baseline score as the covariate

27. Secondary Outcome: Mean Change From Baseline to Month 9 for PAGI-SYM Total Score
Description: as for outcome 24
Time Frame: Baseline and Month 9
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Number analyzed (Participants) | 109 | 292
score on a scale | -1.17 (0.902) | -0.89 (0.903)
Statistical Analysis 1: Comparison: Dexlansoprazole MR 60 mg QD vs Dexlansoprazole MR 90 mg QD; Test type: Superiority or Other; p = 0.005, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Comparisons were made using an ANCOVA model with treatment as the factor and baseline score as the covariate

28. Secondary Outcome: Mean Change From Baseline to Month 12 for PAGI-SYM Total Score
Description: as for outcome 24
Time Frame: Baseline and Month 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Number analyzed (Participants) | 95 | 236
score on a scale | -1.08 (0.915) | -0.95 (0.879)
Statistical Analysis 1: Comparison: Dexlansoprazole MR 60 mg QD vs Dexlansoprazole MR 90 mg QD; Test type: Superiority or Other; p = 0.469, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Comparisons were made using an ANCOVA model with treatment as the factor and baseline score as the covariate

29. Primary Outcome: Changes From Baseline to Final Visit in Antrum Biopsy Results
Description: Normal=normal tissue; Unknown Baseline = Baseline biopsy not available; Abnormal diagnoses include: Reactive Gastropathy, Chronic Gastritis, Intestinal Metaplasia, Reflective Observation Mucosa-Associated Lymphoid Tissue Lymphoma, Other Abnormal.
Time Frame: Baseline and Final Visit (up to 12 months)
Population: All subjects with Final Visit antrum biopsies are included. Each subject is counted only once per tissue type based on the worst diagnosis. Final Visit was the last visit of this study and no more than 14 days post-dosing.
Measure: Number; unit: subjects
Arm/Group | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Number analyzed (Participants) | 102 | 297
subjects
  Normal Baseline to Normal Final Visit | 39 | 114
  Normal Baseline to Abnormal Final Visit | 11 | 61
  Abnormal Baseline to Normal Final Visit | 21 | 47
  Abnormal Baseline to Abnormal Final Visit | 29 | 60
  Unknown Baseline to Normal Final Visit | 1 | 11
  Unknown Baseline to Abnormal Final Visit | 1 | 4

30. Primary Outcome: Changes From Baseline to Final Visit in Fundus Biopsy Results
Description: as for outcome 29
Time Frame: Baseline and Final Visit (up to 12 months)
Population: All subjects with Final Visit fundus biopsies are included. Each subject is counted only once per tissue type based on the worst diagnosis. Final Visit was the last visit of this study and no more than 14 days postdosing.
Measure: Number; unit: subjects
Arm/Group | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Number analyzed (Participants) | 103 | 306
subjects
  Normal Baseline to Normal Final Visit | 55 | 198
  Normal Baseline to Abnormal Final Visit | 8 | 35
  Abnormal Baseline to Normal Final Visit | 17 | 33
  Abnormal Baseline to Abnormal Final Visit | 21 | 35
  Unknown Baseline to Normal Final Visit | 2 | 2
  Unknown Baseline to Abnormal Final Visit | 0 | 3

ADVERSE EVENTS:
Arm/Group | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Serious Adverse Events (participants affected / at risk) | 9 | 21
Other Adverse Events (participants affected / at risk) | 63 | 165
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Neutropenias (Blood and lymphatic system disorders) | 0/153 | 1/438
Inner Ear Signs and Symptoms (Ear and labyrinth disorders) | 0/153 | 1/438
Duodenal and Small Intestinal Stenosis and Obstruction (Gastrointestinal disorders) | 0/153 | 1/438
Pain and Discomfort NEC (General disorders) | 0/153 | 2/438
Cholecystitis and Cholelithiasis (Hepatobiliary disorders) | 1/153 | 2/438
Anaphylactic Responses (Immune system disorders) | 0/153 | 1/438
Abdominal and Gastrointestinal Infections (Infections and infestations) | 2/153 | 0/438
Lower Respiratory Tract and Lung Infections (Infections and infestations) | 1/153 | 0/438
Staphylococcal Infections (Infections and infestations) | 0/153 | 1/438
Upper Respiratory Tract Infections (Infections and infestations) | 1/153 | 0/438
Urinary Tract Infections (Infections and infestations) | 0/153 | 1/438
Lower Limb Fractures and Dislocations (Injury, poisoning and procedural complications) | 0/153 | 1/438
Non-Site Specific Injuries NEC (Injury, poisoning and procedural complications) | 0/153 | 4/438
Non-Site Specific Procedural Complications (Injury, poisoning and procedural complications) | 0/153 | 1/438
Thoracic Cage Fractures and Dislocations (Injury, poisoning and procedural complications) | 0/153 | 1/438
Upper Limb Fractures and Dislocations (Injury, poisoning and procedural complications) | 0/153 | 1/438
Intervertebral Disc Disorders NEC (Musculoskeletal and connective tissue disorders) | 0/153 | 3/438
Joint Related Disorders NEC (Musculoskeletal and connective tissue disorders) | 0/153 | 1/438
B-cell Lymphomas NEC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/153 | 1/438
Leukaemias Acute Myeloid (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/153 | 0/438
Neoplasms Benign Site Unspecified NEC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/153 | 1/438
Renal Neoplasms Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/153 | 1/438
Uterine Neoplasms Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/153 | 0/438
Disturbances in Consciousness NEC (Nervous system disorders) | 1/153 | 1/438
Migraine Headaches (Nervous system disorders) | 1/153 | 0/438
Perception Disturbances (Psychiatric disorders) | 0/153 | 1/438
Renal Lithiasis (Renal and urinary disorders) | 0/153 | 1/438
Bronchospasm and Obstruction (Respiratory, thoracic and mediastinal disorders) | 1/153 | 0/438
Pneumothorax and Pleural Effusions NEC (Respiratory, thoracic and mediastinal disorders) | 0/153 | 1/438
Pulmonary Thrombotic and Embolic Conditions (Respiratory, thoracic and mediastinal disorders) | 0/153 | 1/438
Respiratory Failures (Excl Neonatal) (Respiratory, thoracic and mediastinal disorders) | 1/153 | 0/438
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Diarrhoea (Excl Infective) (Gastrointestinal disorders) | 18/153 | 34/438
Flatulence, Bloating, and Distension (Gastrointestinal disorders) | 6/153 | 26/438
Gastrointestinal and Abdominal Pains (Excl Oral and Throat) (Gastrointestinal disorders) | 10/153 | 47/438
Nausea and Vomiting Symptoms (Gastrointestinal disorders) | 13/153 | 41/438
Upper Respiratory Tract Infections (Infections and infestations) | 22/153 | 59/438
Musculoskeletal and Connective Tissue Signs and Symptoms NEC (Musculoskeletal and connective tissue disorders) | 11/153 | 23/438
Headaches NEC (Nervous system disorders) | 11/153 | 27/438

LIMITATIONS AND CAVEATS:
The incidence of adverse events was considered one of the primary outcome measures of this study. These results are presented in the Adverse Events Section and are not reposted as a separate primary endpoint.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be published prior to publication of a multi-center report submitted for publication within 18 months after conclusion or termination of a study. Results publications will be submitted to sponsor for review 60 days in advance of publication. Sponsor can require removal of confidential information unrelated to study results. Sponsor can embargo a proposed publication for another 60 days to preserve intellectual property.